CLINICAL TRIAL: NCT06461949
Title: A Randomized, 52-Week Treatment Double-Blind, Placebo-Controlled Efficacy and Safety Study of Dupilumab 300 mg Every Other Week After Endoscopic Sinus Surgery in Patients With Allergic Fungal Rhinosinusitis (AFRS) on a Background Therapy With Intranasal Corticosteroid Spray
Brief Title: Study of Dupilumab 300 mg Every Other Week After Endoscopic Sinus Surgery in Patients With Allergic Fungal Rhinosinusitis (AFRS) on a Background Therapy With Intranasal Corticosteroid Spray
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Closed by sponsor, lack of enrollment.
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10001856; 001856-DC
Record Dates: First submitted 2024-06-08; First posted 2024-06-17 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Allergic Fungal Rhinosinusitis (AFRS); Chronic Rhinosinusitis (CRS); Asthma; Nasal Polyps
Keywords: Ethmoid tissue; Intranasal corticosteroids; Nasal polyps; Sinonasal inflammation; Lung Function; Quality of Life
MeSH Terms: conditions — Allergic Fungal Sinusitis; Asthma; Nasal Polyps | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: (Experimental): Treatment: Dupilumab 300 mg administered subcutaneously every two weeks for 52 weeks.
  Interventions: Drug: Dupilumab
- Arm B: (Placebo Comparator): Control: Placebo administered subcutaneously every two weeks for 52 weeks.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Dupilumab (Dupixent) is a human monoclonal antibody administered via subcutaneous injection to treat various conditions such as Chronic Rhinosinusitis with Nasal Polyps, Asthma and Eosinophilic Esophagitis.

SUMMARY:
Background:

Allergic fungal rhinosinusitis (AFRS) is a severe type of sinus infection. People with AFRS develop heavy mucus and growths called polyps that apply pressure to the sinuses and block their breathing. Surgery can remove the polyps, but they often grow back. Researchers want to test an approved drug they believe may help people with AFRS.

Objective:

To test a drug (Dupilumab) in people with AFRS.

Eligibility:

People aged 18 years or older with suspected AFRS who are scheduled to undergo surgery for nasal polyps.

Design:

Participants will have several tests before their surgery. They will have imaging scans of their sinuses. They will have an endoscopic exam: A tube with a camera and a light will be inserted into their sinuses. They may give blood and mucus samples. They will have standard treatment with nasal sprays for 2 to 6 weeks before their surgery.

Excess nasal tissue removed during the surgery will be collected for research. Then they will begin treatment with the study drug.

Dupilumab is injected under the skin. Some participants will receive the study drug. Some will receive a placebo injections. The placebo injections are just like the study drug but contain no medicine. Participants will not know which injections they are getting.

All participants will administer the injections to themselves at home. They will do this every 2 weeks for 1 year after the surgery. They will have a clinic visit 16 weeks after surgery.

Participants will have follow-up for 12 weeks after treatment ends.

DETAILED DESCRIPTION:
Study Description:

Multicenter, randomized, double-blind, placebo-controlled study comparing the efficacy of dupilumab to placebo in allergic fungal rhinosinusitis (AFRS) subjects after sinus surgery on a background treatment with intranasal corticosteroid spray.

Study periods:

The clinical trial consists of 4 periods:

-Run-in period (2 weeks + 4 weeks):

All participants will enter a run-in period of 2-6 weeks receiving saline irrigations and Intranasal Corticosteroids per the treating physician. All oral steroids and antibiotics will be stopped.

-Ethmoid Tissue Collection period (7 days + 4 weeks):

Participants will undergo surgery as scheduled per standard of care. Ethmoid tissue will be collected from all subjects at the time of surgery.

-Randomized treatment (52 weeks +/- 7 days):

Participants will be randomized to one of the following treatments:

* Arm A: dupilumab 300 mg subcutaneous (SC) every two weeks for 52 weeks
* Arm B: placebo given SC every two weeks for 52 weeks

  * Posttreatment period (12 weeks +/- 7 days):

After completing 52 weeks of treatment with IMP (or following early discontinuation of IMP), subjects will be instructed to:

* Return to the study site for the last scheduled visits for physical examination, nasal endoscopy, Nasal Polyps Score (NPS), Patient-Reported Outcomes (PROs)(Sinonasal Outcomes Test-SNOT-22-, and Asthma Control Questionnaire -ACQ-), FEV1 measurement in those with asthma, and safety.
* Continue on stable dose of INCS spray during the posttreatment period.
* Report any adverse event (AE).

Co-Primary Objectives:

* Determine the efficacy of dupilumab in controlling sinonasal inflammation and preventing nasal polyp recurrence after complete sinus surgery for AFRS as measured by change in the mLK score.
* Evaluate the effect of dupilumab on oral corticosteroid utilization following complete sinus surgery for AFRS.

Secondary Objectives:

To evaluate the effect of dupilumab on:

* Prevention of revision surgery for AFRS
* Secondary objective measures of sinonasal inflammation following sinus surgery using NPS and LMS.
* Lower airway dysfunction following sinus surgery in the subgroup of participants with asthma (approximately 25%)
* Upper and lower airway, disease-specific, health-related quality of life, as measured by ACQ and SNOT-22
* Reducing utilization of rescue medications for acute exacerbations of CRS following sinus surgery

Primary Endpoints:

Change from baseline at 52 weeks both within and between treatment and placebo arms:

* Endoscopic modified Lund-Kennedy (mLK) score
* Incidence of oral corticosteroid utilization per participant

Secondary Endpoints:

Change from baseline at 52 weeks both within and between treatment and placebo arms:

* Prevalence of revision sinus surgery for recurrent nasal polyps, and comparison of survival curves
* Endoscopic nasal polyp score (NPS)
* CT generated Lund-McKay score
* Spirometry (for participants with comorbid asthma)
* 22-item sinonasal outcomes test (SNOT-22)
* Asthma Control Questionnaire (ACQ)
* Prevalence of oral / topical corticosteroid utilization per treatment cohort
* Incidence of oral / topical antibiotic utilization per subject
* Prevalence of oral / topical antibiotic utilization per treatment cohort

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants are eligible for study participation if all inclusion and no exclusion criteria are met. Non- English-speaking people will be included if they fulfill the criteria. In order to be eligible to participate in this study, an individual must meet all of the following criteria:

Informed consent

* Participants must be capable of giving signed informed consent as listed in the informed consent form (ICF) and this protocol.
* ICF must be signed and dated prior to study specific procedures. Informed consent process is described further below.

Age

-Participants aged >=18 years at the time of signing the ICF.

Types of subject and disease characteristics

* Participants with nasal polyps in the setting of suspected AFRS and electing to undergo comprehensive sinus surgery per established criteria.

  * Diagnosis of nasal polyps by consensus criteria.
  * Failure of appropriate medical therapy, including topical intranasal corticosteroid (spray or irrigation) > 8 weeks duration, systemic corticosteroid trial of 1-3 weeks duration and nasal saline irrigation of > 4 weeks duration.
  * A minimum SNOT-22 score of 20 at time of enrollment.
  * A minimum CT Lund-MacKay score of > 1 at time of enrollment.
* Suspected AFRS based on Bent and Kuhn criteria

  * Participants must meet 3/5 criteria at time of enrollment

    * Environmental atopy by skin or serum testing
    * Nasal polyposis
    * Characteristic CT findings
    * Eosinophilic mucous
    * Fungal identification on histopathology
  * Participants must meet 5/5 criteria at time of randomization.

Enrolled subjects are expected to undergo SoC allergy testing and sinus surgery prior to randomization. This will complete evaluation for suspected AFRS, thus enabling further study participation. Allergy testing & sinus surgery, in addition to other SoC items, will be done per clinical guidelines at the treating institution and will not be covered in this protocol.

Sinus Surgery

-All study participants will have met criteria for sinus surgery and undergo a comprehensive procedure prior to randomization. The procedure will not be assigned and will be completed per SoC at the treating institution for the management of nasal polyps in suspected AFRS.

Reproduction

* Negative urine pregnancy test will be required at enrollment and study visits 3, 4, 5 and 6, throughout the treatment period for participants of childbearing potential (i.e., post-pubescent, premenopausal females).
* Persons of childbearing potential must use an effective form of birth control (confirmed by the Investigator) e.g., total sexual abstinence, vasectomized sexual partner, tubal occlusion, intrauterine device or levonorgestrel Intrauterine system, Depo-Provera injections, oral contraceptive, Evra Patch, or Nuvaring. Women of childbearing potential must agree to use a highly effective method of birth control, as defined above, from enrollment, throughout the study duration and for 12 weeks after the last dose of IMP.
* To protect against possible side effects, men should not get a sexual partner pregnant while taking the study drug and for 12 weeks after the last dose. Men should agree on a method of birth control to use throughout the study.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

Medical Conditions:

* Participants who have undergone nasal or sinus surgery within 3 months prior to enrollment.
* Participants with conditions or comorbid disease findings that preclude nasal endoscopy for evaluation of primary outcome, such as:

  * Current rhinitis medicamentosa
  * Nasal cavity tumors
  * Occlusive septal deviation following surgery
* Clinically important comorbidities that may confound interpretation of clinical efficacy, including:

  * Aspirin-exacerbated respiratory disease
  * Cystic fibrosis
  * Primary ciliary dyskinesia
  * Hereditary Hemorrhagic Telangiectasia
  * Antrochoanal polyposis
  * Non-asthma eosinophilic disease, such as bronchopulmonary aspergillosis, eosinophilic granulomatosis with polyangiitis, hypereosinophilic syndrome
  * Granulomatosis with polyangiitis
  * Any corticosteroid dependent condition
* A comorbid health disorder that is not medically controlled in the opinion of the Investigator, and has the potential to:

  * Affect the safety of the subject throughout the study
  * Impede the subject s ability to complete the duration of the study
  * Influence the primary or secondary outcomes of the study
* Participant experiencing a symptomatic asthma exacerbation requiring systemic corticosteroids or hospitalization (>24 hours) within 4 weeks of randomization.
* Infection requiring systemic antibiotics within 4 weeks of randomization.

  --Parenteral and/or oral antibiotics associated with surgery are allowed
* Medical contraindication to receiving dupilumab:

  * Known hypersensitivity to dupilumab or any of its excipients
  * Live vaccine administration within 30 days of randomization or during study period
  * Known helminth infection.
* Unable to tolerate sinonasal irrigations.
* Pregnancy, current lactation, or lack of effective contraception plan, as determined by the site investigator.

Prior Concomitant Therapy

* Initiation of allergen immunotherapy within 3 months prior to randomization or a plan to begin therapy or change its dose during the study period.
* Immunosuppressive medication within 3 months prior to randomization and during the study period from randomization through EOS.
* Receipt of any marketed or investigational biologic products (monoclonal or polyclonal antibody) within 6 months or 5 half-lives, whichever is longer, prior to randomization during the study period.
* Previous use of dupilumab.
* Receipt of immunoglobulin or blood products within 30 days prior to randomization.
* Receipt of any investigational drug within 30 days or 5 half-lives, whichever is longer prior to randomization.
* Scheduled systemic corticosteroid treatment during the study period:

  --Standardized corticosteroid taper associated with planned surgery is allowed.
* Receipt of leukotriene antagonists or modifiers for participants who were not on a stable dose for > 30 days prior to randomization

Prior/concurrent clinical study experience

-Concurrent enrollment in another investigational drug trial during the study period.

Other Exclusions

* Participant involvement in the planning or conduct of the study.
* Investigator assessment that the subject is unlikely to comply with study procedures.
* Prior randomization in the present study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Efficacy of Dupilumab | Change from baseline at 52 weeks
  -Control of sinonasal inflammation.-Prevention of nasal polyp recurrence after complete sinus surgery for AFRS.-Measured by change in the modified Lund-Kennedy (mLK) score.

SECONDARY OUTCOMES:
Effect of Dupilumab on Oral Corticosteroid Utilization | Change from baseline at 52 weeks
  Reduction in the use of oral corticosteroids following complete sinus surgery for AFRS.
Prevention of Revision Surgery for AFRS | Change from baseline at 52 weeks
  Assessment of the need for additional surgery due to recurrent nasal polyps.
Secondary Objective Measures of Sinonasal Inflammation | Change from baseline at 52 weeks
  Changes in nasal polyp score (NPS) and CT-generated Lund-McKay score (LMS).
Lower Airway Dysfunction in Participants with Asthma | Change from baseline at 52 weeks
  Spirometry measurements and other assessments in approximately 25% of participants with asthma
Health-Related Quality of Life | Change from baseline at 52 weeks
  Upper and lower airway disease-specific quality of life measured by the Asthma Control Questionnaire (ACQ) and the Sinonasal Outcomes Test (SNOT-22).
Utilization of Rescue Medications | Change from baseline at 52 weeks
  Reduction in the use of rescue medications for acute exacerbations of chronic rhinosinusitis (CRS) following sinus surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Levy, M.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)

IPD SHARING:
Plan to Share IPD: Yes
.Research Data for Statistical Analysis and Scientific Reporting will be shared. All participant data will be de-identified. Participants will be identified only by a unique study identification number.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Post study completion and as determined by NIDCD staff.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001856-DC.html